CLINICAL TRIAL: NCT06080880
Title: Ondanstron Weekly vs Every 3 Weeks for Prevention of Nausea and Vomiting Induced by Chemotherapy Combined With PD-1 Blockade：an Randomized Clinical Trial
Brief Title: Ondanstron Weekly vs Every 3 Weeks for Prevention of Nausea and Vomiting Induced by Chemotherapy Combined With PD-1 Blockade
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, Director of the department of Radiotherapy Oncology, Hubei Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-143-001
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Nausea With Vomiting Chemotherapy-Induced
Keywords: Chemotherapy-induced nausea and vomiting; PD-1 blockade; Ondanstron
MeSH Terms: conditions — Vomiting | interventions — Aprepitant; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron every 3 weeks combined with aprepitant and dexamethasone (Experimental)
  Interventions: Drug: Ondansetron every 3 weeks; Drug: Aprepitant; Drug: Dexamethasone
- Ondansetron weekly combined with aprepitant and dexamethasone (Experimental)
  Interventions: Drug: Aprepitant; Drug: Dexamethasone; Drug: Ondansetron weekly

INTERVENTIONS:
Drug: Ondansetron every 3 weeks — Ondansetron, Po, 24mg/d, 3 days' application every 3 weeks
  Arms: Ondansetron every 3 weeks combined with aprepitant and dexamethasone
Drug: Aprepitant — aprepitant, Po, 125mg/d, 1day' application every 3 weeks
Drug: Dexamethasone — dexamethasone, iv, 10mg/d, 1day' application every 3 weeks
Drug: Ondansetron weekly — Ondansetron, Po, 24mg/d, 3 days' application weekly
  Arms: Ondansetron weekly combined with aprepitant and dexamethasone

SUMMARY:
The aim of this randomized study is to compare the efficacy and safety of ondanstron weekly with every 3 weeks for the prevention of nausea and vomiting induced by chemotherapy combined with PD-1 blockade.

DETAILED DESCRIPTION:
Nausea and vomiting have become the most common and intolerant adverse events in patients receiving chemotherapy, which cause substantial impairments in human functions and quality of life. In some serious cases, patients refused further treatment and lead to disruption of the course of treatment.

For highly emetogenic chemotherapy(HEC), a standard triple therapy including 5-hydroxytryptamine-3 receptor antagonist(5-HT3RA), neurokinin-1 receptor antagonist(NK-1RA) plus corticosteriod. Recently, a few trials have achieved success in reduction of post-discharge application of corticosteriod based on the standard triple therapy, which offered new insights to update the current therapeutic regimens.

Although the emetogenicity of PD-1 blockade seems to be slighter than HEC, previous studies have reported gastrointestinal immune-related adverse events(GI-IrAE) in patients treated with PD-1 blockade, of which 55% of the participants suffered nausea and vomiting. Noteworthy, recently researchers highlight the importance of prevention and control of nausea more than that of vomiting in terms with chemotherapy-induced nausea and vomiting.

Therefore, the investigators initiated this study to compare the efficacy and safety of ondanstron weekly with every 3 weeks for the prevention of nausea and vomiting induced by chemotherapy combined with PD-1 blockade, which may provide new insights for fully prevention and control compare the efficacy and safety of ondanstron weekly with every 3 weeks for the prevention of nausea and vomiting induced by chemotherapy combined with PD-1 blockade in aimed population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender limit;
2. Pathologically or cytologically confirmed malignant solid tumors;
3. Scheduled to receive cisplatin-based chemotherapy combined with PD-1 blockade；
4. TPS > 1 %(PD-1);
5. Adequate hematological function (leucocyte count ≥ 4000/μL [to convert to ×109/L,multiply by 0.001], hemoglobin ≥ 9.00 g/dL [to convert to grams per liter, multiply by 10], and platelet count ≥ 100 × 103/μL [to convert to ×109/L, multiply by 1]);
6. Hepatic function (alanine aminotransferase and aspartate aminotransferase ≤ 2.0 times the upper limit of the reference ranges), and renal function (creatinine clearance ≥ 60 mL/min/1.73 m2 [to convert to millimeters per second per meter-squared, multiply by 0.0167])；
7. Estimated survival time > 6 months；
8. ECOG 0-1 points；
9. Participants being informed and signed written consents.

Exclusion Criteria:

1. Nausea or vomiting caused by reasons except for chemotherapy and PD-1 blockade;
2. Participants with other malignant tumors history previously;
3. Inability to read, comprehend, and finish questionnaires;
4. Allergic to the drugs included in this study.
5. Administered drugs with antiemetic activity within the 24 hours before receiving the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Complete response(CR) rate | Up to 6 weeks
  Defined as no emesis and no rescue therapy

SECONDARY OUTCOMES:
The proportion of patients with sustained no emesis, sustained no nausea, sustained no significant nausea, and the mean time to first emetic episode. | Assessed every week
  The proportion of patients with sustained no emesis, sustained no nausea, sustained no significant nausea (defined as no or mild nausea), and the mean time to first emetic episode.

CONTACTS AND LOCATIONS:
Overall Officials: Guang Han, MD, Principal Investigator — Hubei Cancer Hospital, Wuhan, HuBei, China, 430079
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No